CLINICAL TRIAL: NCT05274412
Title: Clinical Efficacy of Hypotension Prediction Index Based Perioperative Protocolized Hemodynamic Management in Geriatric Orthopedic Surgery
Brief Title: Hypotension Prediction Index Based Perioperative Protocolized Hemodynamic Management in Geriatric Orthopedic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 202112163RIND
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2022-03

CONDITIONS: Orthopedic Disorder; Hemodynamic Instability
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Participants in this group will receive protocolized hemodynamic management based on advanced hemodynamic monitoring and dynamic parameters.Keep pulse pressure variation >12%; keep cardiac index >2L/min/cm^2; keep mean arterial pressure > 65mmHg.
  Interventions: Other: ordinary goal-directed hemodynamic therapy
- HPI group (Experimental): Participants in this group will receive protocolized hemodynamic management based on advanced hemodynamic monitoring, hypotension prediction index (HPI), and dynamic parameters.Keep HPI <85; pulse pressure variation >12%; keep cardiac index >2L/min/cm^2; keep mean arterial pressure > 65mmHg.
  Interventions: Other: hypotension prediction index(HPI)

INTERVENTIONS:
Other: hypotension prediction index(HPI) — Implementing hypotension prediction index (HPI) in perioperative goal-directed hemodynamic therapy. Keep HPI < 85; pulse pressure variation >12%; keep cardiac index >2L/min/cm^2; keep mean arterial pressure > 65mmHg.
  Arms: HPI group
Other: ordinary goal-directed hemodynamic therapy — Keep pulse pressure variation >12%; keep cardiac index >2L/min/cm^2; keep mean arterial pressure > 65mmHg.
  Arms: Control group

SUMMARY:
Blood pressure optimization has been considered as a crucial factor to avoid perioperative vital organ hypoperfusion, and perioperative hypotension has been addressed as a risk factor for complications and adverse clinical outcomes.

Hypotension prediction index (HPI) is an novel machine-learning derived parameters, and was developed to predict the risk of future hypotension.Series of clinical studies have verified its clinical efficacy in avoiding perioperative hypotension.

Major orthopedic surgeries, such as spine surgery, joint surgery, long bone fracture surgery, are quite common in elder people, who are vulnerable to perioperative adverse outcomes.Thus the investigator design this study to testify the clinical efficacy of implementing HPI in perioperative goal-directed hemodynamic therapy in elder patients receiving major orthopedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* adults elder or equal to 60 years old receiving scheduled orthopedic surgery

Exclusion Criteria:

* Patients with a history of arrhythmia, congestive heart failure, preoperative neurocognitive disorder, cerebrovascular event, chronic obstructive pulmonary disease, chronic kidney disease, ongoing infectious disease, will be excluded.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Perioperative acute kidney injury | 24 hours
  Acute kidney injury will be assessed according to the KDIGO guideline. Serum creatinine will be examined on the day before surgery and postoperative day 1.

OTHER OUTCOMES:
perioperative neurocognitive disorder | 30 day
  Taiwan version of quick mild cognitive impairment(Qmci) test will be used to identify perioperative neurocognitive disorder

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Tse Lee, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monk TG, Bronsert MR, Henderson WG, Mangione MP, Sum-Ping ST, Bentt DR, Nguyen JD, Richman JS, Meguid RA, Hammermeister KE. Association between Intraoperative Hypotension and Hypertension and 30-day Postoperative Mortality in Noncardiac Surgery. Anesthesiology. 2015 Aug;123(2):307-19. doi: 10.1097/ALN.0000000000000756. PMID 26083768
- [Background] Wesselink EM, Kappen TH, Torn HM, Slooter AJC, van Klei WA. Intraoperative hypotension and the risk of postoperative adverse outcomes: a systematic review. Br J Anaesth. 2018 Oct;121(4):706-721. doi: 10.1016/j.bja.2018.04.036. Epub 2018 Jun 20. PMID 30236233
- [Result] Hatib F, Jian Z, Buddi S, Lee C, Settels J, Sibert K, Rinehart J, Cannesson M. Machine-learning Algorithm to Predict Hypotension Based on High-fidelity Arterial Pressure Waveform Analysis. Anesthesiology. 2018 Oct;129(4):663-674. doi: 10.1097/ALN.0000000000002300. PMID 29894315
- [Result] Wijnberge M, Geerts BF, Hol L, Lemmers N, Mulder MP, Berge P, Schenk J, Terwindt LE, Hollmann MW, Vlaar AP, Veelo DP. Effect of a Machine Learning-Derived Early Warning System for Intraoperative Hypotension vs Standard Care on Depth and Duration of Intraoperative Hypotension During Elective Noncardiac Surgery: The HYPE Randomized Clinical Trial. JAMA. 2020 Mar 17;323(11):1052-1060. doi: 10.1001/jama.2020.0592. PMID 32065827